CLINICAL TRIAL: NCT00724386
Title: A Phase I Study of Concomitant Chemoradiotherapy With Weekly Paclitaxel and Vinorelbine With Filgrastim Granulocyte Colony Stimulating Factor (GCSF) Support in Patients With Advanced Breast Cancer
Brief Title: Concomitant Chemoradiotherapy With Weekly Paclitaxel and Vinorelbine and Granulocyte Colony Stimulating Factor (GCSF) Support in Patients With Advanced Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCIRB 9849
Record Dates: First submitted 2008-07-25; First posted 2008-07-29 (Estimated); Last update posted 2014-03-07 (Estimated); Status verified 2014-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Paclitaxel; Vinorelbine; Filgrastim; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Paclitaxel — 1-hour IV infusion once weekly for 12 to 14 weeks
  Other Names: Taxol
Drug: Vinorelbine — escalating doses administered intravenously over 6-10 minutes for 12-14 weeks
  Other Names: Navelbine
Drug: Filgrastim — daily injections for 6 days beginning on day 2 of second week on study and then every other week (weeks 2, 4, 6, 8, 12).
  For the final dose cohort, administration on chemotherapy only weeks, only if dose reduction or dose delay required by subject
Radiation: Radiation — Radiotherapy for 5 consecutive days every other week (weeks 1, 3, 5, 7, 9, 11, 13)starting on same day as first dose of protocol chemotherapy

SUMMARY:
The goal of this study is to determine the feasibility based on toxicity and response rate of giving paclitaxel weekly with concomitant every-other week radiotherapy to limit skin toxicity. This study will also seek to determine the maximally tolerated dose of Navelbine added to this combination when followed by Filgrastim and the dose-limiting toxicities of this regimen.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the male or female breast (male or female) with gross, uncontrolled, unresectable breast and/or chest wall disease including:

  1. patients with locally advanced unresectable stage IIIa or IIIb;
  2. patients with locally recurrent (including locoregional lymph nodes) disease for which curative surgery is not thought possible
  3. patients with metastatic disease AND uncontrolled locoregional disease are eligible.
* Prior chemotherapy allowed, except for nitrosoureas and mitomycin chemotherapy or high dose chemotherapy with marrow or stem cell rescue.
* Prior palliative radiation to sites of metastases allowed (i.e. bone, brain, lung)
* 4 weeks since any prior treatments (excluding hormonal therapy). Concurrent hormonal therapy is not allowed.
* Aged 18 years or older
* CALGB performance status of 0 - 2
* Life expectance of at least 12 weeks
* Initial Laboratory Data:

  * ANC Count > 1500/mm3
  * Platelet Count > 100,000/mm3
  * Creatine ≤ 2.0 mg/dl
  * Bilirubin ≤ 1.5 mg/dl
  * ALT (SGPT) ≤ 3 times the upper limit of normal
* Signed informed consent

Exclusion Criteria:

* Prior breast or chest wall radiation is not allowed unless the proposed site radiation port does not overlap with prior ports
* Subjects must not be pregnant (females able to have children must have negative pregnancy test and agree to use adequate contraception)
* Patients with a documented hypersensitivity to E.coli derived proteins are excluded.
* No other serious medical condition such as uncontrolled infection that in the opinion of the investigators places patient at undue risk for study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 1999-06; Primary Completion 2005-10 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
feasibility of administering study therapy to limit skin toxicity | 4 weeks
dose-limiting toxicity | 4 weeks

SECONDARY OUTCOMES:
response | 14 weeks
time to progression
overall survival
Bcl-2 detection by immunohistochemistry | 14 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- University of Chicago, Chicago, Illinois, United States